CLINICAL TRIAL: NCT02946541
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial to Investigate the Efficacy and Safety of Evogliptin After Oral Administration in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Diet and Exercise
Brief Title: A Clinical Trial to Investigate the Efficacy and Safety of Evogliptin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1229_DMM_III
Record Dates: First submitted 2014-02-23; First posted 2016-10-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DA-1229; evogliptin; DPP-IV inhibitor; Suganon; DPP-4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- evogliptin 5mg (Experimental): evogliptin 5mg QD
  Interventions: Drug: evogliptin 5mg
- placebo (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: evogliptin 5mg — evogliptin 5mg, QD
  Other Names: DA-1229; Suganon
  Arms: evogliptin 5mg
Drug: Placebo — Placebo, QD
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase III clinical trial to investigate the efficacy and safety of evogliptin after oral administration in patients with type 2 diabetes who have inadequate glycemic control on diet and exercise.

DETAILED DESCRIPTION:
1. Evogliptin 5mg Group: Administration with Evogliptin 5mg for 0-52 weeks.
2. Placebo Group: Administration with Placebo for 0-24 weeks, and with Evogliptin 5mg for 24-52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 6.5%≤HbA1c≤10.0% at screening
* Subjects untreated with oral hypoglycemic agents within 6 weeks prior to screening
* Subjects with 6.5%≤HbA1c≤10.0% at Visit 2
* Subjects with 20kg/m2≤BMI≤40kg/m2 at screening

Exclusion Criteria:

* Subjects with fasting plasma glucose≥270mg/dL at screening
* Patients with type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* Subjects with history of myocardial infarction, cerebral infarction within 6 months prior to screening
* Subjects with ALT and AST 2.5 times or higher than upper normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline at 24 weeks
  unit: %

SECONDARY OUTCOMES:
fasting plasma glucose | Change from baseline at 24 weeks
  unit: mg/dL
HbA1c response rate | Change from baseline at 24 weeks
  unit: %

CONTACTS AND LOCATIONS:
Overall Officials: Doo Man Kim, M.D., Ph.D., Principal Investigator — Kangdong Sacred Heart Hospital
Locations (1):
- Kangdong Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No